CLINICAL TRIAL: NCT01598207
Title: The Effects of Cannabinoid on Patients With Non-GERD Related Non Cardiac Chest Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yehudith Assouline-Dayan (Other)
Responsible Party: Sponsor-Investigator, Yehudith Assouline-Dayan, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201003768
Record Dates: First submitted 2012-05-10; First posted 2012-05-15 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Marinol (Experimental)
  Interventions: Drug: Marinol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Marinol — 5mg BID, orally for 1 month
  Arms: Marinol
Drug: Placebo — 5mg BID, orally for 1 month
  Arms: Placebo

SUMMARY:
Background: Noncardiac chest pain (NCCP) affects 200,000 new cases annually in USA. It is associated with poor quality of life and high health care expenditure of 8 Billion Dollars a year.

Gastroesophageal Reflux Disease(GERD), esophageal motility disorders, and psychological issues may cause NCCP.

The mechanism(s) for pain continue to be explored and include central and peripheral hypersensitivity, and mechanophysical abnormalities. Treatment of NCCP has focused on relieving visceral hypersensitivity through pain modulators, such as tricyclics, trazodone, or adenosine receptor antagonist, theophylline. Typically, only 40-50 % respond and clearly there is a large unmet therapeutic need.

Cannabis is felt to be beneficial for vomiting, diarrhea and intestinal pain. The main component of Cannabis acts through specific receptors, that are located primarily on central and peripheral neurons (including the enteric nervous system) and myenteric plexus where they modulate neurotransmitter release. Activation of these receptors reduces excitatory enteric transmission and may improve esophageal hyperreactivity and hypersensitivity, the hallmarks of NCCP.

STUDY PROTOCOL: The investigators will randomize 40 subjects with non-cardiac, non-reflux chest pain to receive dronabinol (5 mg Bid), or placebo for 4 weeks. Chest pain symptoms and esophageal sensorimotor properties will be assessed at baseline and at 4 weeks using symptom diary and impedance planimetry. The primary outcome measure will be the frequency of chest pain episodes. Secondary outcome measures include improvement in esophageal sensory thresholds, reduced reactive contractions, frequency, amplitude, area under the curve, and global improvement of symptoms.

HYPOTHESIS: Cannabinoids decrease esophageal hypersensitivity and ameliorate chest pain in NCCP patients, when compared to placebo.

AIM: To perform a randomized double blind study to investigate the effects of Dronabinol, a CB1 and CB2 agonist, in the treatment of patients with NCCP and examine its mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Ages 18-75 years
* Non-GERD related Non cardiac chest pain (Evaluated previously with an EGD, Esophageal manometry, and 24 Hour ambulatory pH study)
* At least one episode of chest pain a week in the past month
* Previous negative cardiac evaluation (EKG ± Non invasive stress test ± Coronary angiogram)

Exclusion Criteria:

* Subjects requiring narcotics or other pain medications
* Subjects with known esophagitis, Barrett's esophagus or peptic stricture on endoscopy
* Subjects with previous upper gastrointestinal surgery
* Pregnancy
* Subjects with Diabetes, neuromuscular disorders, or other severe co-morbidities (Cardiovascular, respiratory, renal, hepatic, hematologic, endocrine, neurologic, and psychiatric)
* Subjects with upper airway symptoms (such as hoarseness, wheezing or laryngospasm)
* Medications such as baclofen, H2 blockers, PPI, sucralfate and prokinetics.
* Known history of substance abuse
* Nursing mothers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Reichenbach ZW, Sloan J, Rizvi-Toner A, Bayman L, Valestin J, Schey R. A 4-week pilot study with the cannabinoid receptor agonist dronabinol and its effect on metabolic parameters in a randomized trial. Clin Ther. 2015 Oct 1;37(10):2267-74. doi: 10.1016/j.clinthera.2015.07.023. Epub 2015 Aug 14. PMID 26283236

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Marinol | Placebo
Started | 7 | 6
Completed | 6 | 6
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Marinol | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Chest Pain Episodes
Description: Number of people still experiencing the same amount of chest pain during treatment than previously without
Time Frame: Baseline and 1 month
Measure: Number; unit: participants
Arm/Group | Marinol | Placebo
Number analyzed (Participants) | 6 | 6
participants | 1 | 3

2. Secondary Outcome: Frequency of Chest Pain in Treatment Group vs Baseline
Description: Total (intensity (0(none) - 3(severe) + duration (0(none) - 3(longer than 30 mins)) at end of 1 month treatment; higher represents worse outcome; the total score ranges from 0 to 6 and is the sum of the intensity and duration
Time Frame: 1 month
Population: 1 participant in placebo did not have this information completed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Marinol | Placebo
Number analyzed (Participants) | 6 | 5
units on a scale | 1.87 (2.58) | 1.8 (1.64)

3. Secondary Outcome: Intensity of Chest Pain Episodes
Description: Intensity (0(none) - 3(severe)) at baseline vs 1 month for chest pain episodes; higher represents worse outcome; multiple chest pain totals are averaged
Time Frame: Baseline and 1 month
Population: 1 participant in placebo did not have this information completed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Marinol | Placebo
Number analyzed (Participants) | 6 | 5
units on a scale
  Baseline | 1.33 (0.82) | 0.6 (0.89)
  1 Month | 0.67 (1.03) | 0.8 (0.84)

4. Secondary Outcome: Sensory Thresholds for First Sensation
Description: This is determined by the Esophageal Balloon Distension Test; range 0-65 mmHg
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Marinol | Placebo
Number analyzed (Participants) | 6 | 6
mmHg | 2 (.125) | 2.7 (.103)

5. Secondary Outcome: Duration of Chest Pain Episodes
Description: 0 - is none and 3 is longer than 30 mins; higher values is worst outcome; chest pain totals are averaged
Time Frame: Baseline vs 1 month
Population: 1 participant in placebo did not have this information completed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Marinol | Placebo
Number analyzed (Participants) | 6 | 5
units on a scale
  Baseline | 1.83 (1.17) | 1 (1.55)
  1 Month | 1.2 (1.64) | 1 (1)

6. Secondary Outcome: Sensory Thresholds for Discomfort
Description: When participants felt pain at earliest pressure; range 0-65 mmHg
Time Frame: Baseline and 1 month
Population: 1 participant in marinol and 1 participant in placebo did not have this information completed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Marinol | Placebo
Number analyzed (Participants) | 5 | 5
mmHg
  Baseline | 6 (5.48) | 5 (5)
  1 Month | 8 (13.04) | 2 (4.47)

7. Secondary Outcome: Sensory Thresholds for Pain
Description: When highest amount of pain was felt; range is 0-65 mmHg
Time Frame: Baseline and 1 month
Population: 1 participant in marinol and 1 participant in placebo did not have this information completed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Marinol | Placebo
Number analyzed (Participants) | 5 | 5
mmHg
  Baseline | 42 (16.81) | 53 (9.75)
  1 Month | 47 (16.8) | 51 (15.17)

ADVERSE EVENTS:
Arm/Group | Marinol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 1/7 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Marinol (N=7) | Placebo (N=6)
Viral Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No